CLINICAL TRIAL: NCT05550246
Title: Identifying Sleep Apnea Patients That Best Respond to Atomoxetine Plus Oxybutynin Therapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Scott Aaron Sands, Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022P001544
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Atomoxetine Hydrochloride; oxybutynin

STUDY DESIGN:
Masking Description: Participants and outcome assessors will be blinded to physiological predicted responder status
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AtoOxy Predicted Responders (Experimental): Participants will take Atomoxetine (80mg) and Oxybutynin (5mg) before bedtime for 3 nights. Half doses will be given on the first night.
  Interventions: Drug: Atomoxetine; Drug: Oxybutynin
- AtoOxy Predicted Nonresponders (Experimental): Participants will take Atomoxetine (80mg) and Oxybutynin (5mg) before bedtime for 3 nights. Half doses will be given on the first night.
  Interventions: Drug: Atomoxetine; Drug: Oxybutynin

INTERVENTIONS:
Drug: Atomoxetine — Treatment given for 3 nights
Drug: Oxybutynin — Treatment given for 3 nights

SUMMARY:
Atomoxetine-plus-oxybutynin therapy (AtoOxy) has been shown to substantially reduce obstructive sleep apnea severity (OSA) in about half of patients. Here, the investigators will study which patients respond meaningfully to therapy using pathophysiological traits measured at baseline sleep studies.

DETAILED DESCRIPTION:
The primary goal of the current study is to test the central hypothesis that therapeutic efficacy of AtoOxy depends on underlying patient pathophysiology.

Aim 1 - Advanced analysis of clinical polysomnography will be used to estimate the OSA traits and classify patients as 'predicted responders' or 'predicted nonresponders'. Investigators will prospectively test whether AtoOxy efficacy is greater in predicted responders.

Aim 2 - Pooling preliminary and prospective data, investigators will test the hypotheses that the following pathophysiological traits are associated with, and therefore predict, greater efficacy: less-severe upper airway collapsibility (less improvement needed to re-establish airflow), lower loop gain (less severe ventilatory control instability), higher arousal threshold (greater scope for muscle activation without arousal), and greater upper airway muscle compensation (functional muscle reflex apparatus).

Aim 3 - Investigators will test the hypothesis that treatment efficacy will be greater in patients with tongue-related upper airway obstruction per previous drug-induced sleep endoscopy results (anterior-posterior collapse patterns).

ELIGIBILITY:
Inclusion Criteria:

* Suspected or diagnosed OSA
* Recent drug induced sleep endoscopy results available (performed as part of routine clinical care).

Exclusion Criteria:

* Any uncontrolled medical condition
* Current use of the medications under investigation
* Use of medications expected to stimulate or depress respiration (including opioids, barbiturates, doxapram, almitrine, theophylline, 4-hydroxybutanoic acid).
* Current use of hypnotic medications (trazodone, eszopiclone, benzodiazepines).
* Current use of SNRIs/SSRIs or anticholinergic medications.
* Conditions likely to affect obstructive sleep apnea physiology: neuromuscular disease or other major neurological disorder, heart failure (also below), or any other unstable major medical condition.
* Respiratory disorders other than sleep disordered breathing: chronic hypoventilation/hypoxemia (awake SaO2 < 92% by oximetry) due to chronic obstructive pulmonary disease or other respiratory conditions.
* Other sleep disorders: periodic limb movements, narcolepsy, or parasomnias.
* Contraindications for atomoxetine and oxybutynin, including:

  * hypersensitivity to atomoxetine or oxybutynin (angioedema or urticaria)
  * pheochromocytoma
  * use of monoamine oxidase inhibitors
  * benign prostatic hypertrophy, urinary retention
  * untreated narrow angle glaucoma
  * bipolar disorder, mania, psychosis
  * history of major depressive disorder (age<24).
  * history of attempted suicide or suicidal ideation within one year prior to screening
  * clinically significant constipation, gastric retention
  * pre-existing seizure disorders
  * clinically-significant kidney disorders (eGFR<60 ml/min/1.73m2)
  * clinically-significant liver disorders
  * clinically-significant cardiovascular conditions
  * moderate-to-severe hypertension (SBP>180 mmHg or DBP>110 mmHg measured at baseline; average of evening and morning measures*)
  * cardiomyopathy (LVEF<50%) or heart failure
  * advanced atherosclerosis
  * history of cerebrovascular events
  * history of cardiac arrhythmias e.g., atrial fibrillation, QT prolongation
  * other serious cardiac conditions that would raise the consequences of an increase in blood pressure or heart rate
  * myasthenia gravis
* Claustrophobia
* Pregnancy or nursing

  n.b. Development of new hypertension that is recognized on the final day of study medications during outcomes collection will not be used as stopping criteria for discontinuing outcomes collection.

Participants that are sexually active and able to become pregnant must agree to use birth control for the entire study.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypopnea index (AHI) | 3 days
  Apneas and hypopneas per hour (3% desat and/or arousal), % change from baseline

SECONDARY OUTCOMES:
Hypoxic Burden | 3 days
  Desaturation area under curve × event frequency
Arousal Index | 3 days
  Number of arousals per hour (>=3-sec), % change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Sands, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be available to researchers who provide a methodologically sound proposal.
  All IPD collected during the study will be available after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately after publication. No end date.
Access Criteria: 1-page proposals should be directed to Dr. Scott Sands (sasands@bwh.harvard.edu). To gain access, requestors will be asked to sign a data use agreement.